CLINICAL TRIAL: NCT05458869
Title: Qualitative Study of HPV Self-Collection Experience and Cervical Cancer Screening in Patients With a History of Sexual Trauma
Brief Title: Evaluating the Human Papillomavirus Self-Collection Experience in Individuals Who Have Experienced Sexual Trauma
Status: Completed | Type: Observational
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Oregon Health and Science University (Other); Robert Wood Johnson Foundation (Other)
Responsible Party: Principal Investigator, Amanda Bruegl, MD, Principal Investigator, OHSU Knight Cancer Institute
Other Study IDs: STUDY00024429; NCI-2022-05454 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00024429 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2022-07-12; First posted 2022-07-14 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Cervical Carcinoma; Human Papillomavirus Infection
MeSH Terms: conditions — Uterine Cervical Neoplasms; Papillomavirus Infections | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (survey, HPV self-collection, interview): Participants complete a survey, use an HPV self-collection kit, and attend an interview over 30 minutes.
  Interventions: Procedure: HPV Self-Collection; Other: Interview; Other: Survey Administration

INTERVENTIONS:
Procedure: HPV Self-Collection — Use HPV self-collection kit
  Other Names: At-home HPV Self Collection; HPV Self Collection; Human Papillomavirus Self-Collection
Other: Interview — Attend interview
Other: Survey Administration — Complete surveys

SUMMARY:
This study explores the human papillomavirus (HPV) self-collection experience among individuals with a history of sexual trauma. Cervical cancer is the fourth most common cancer in women worldwide and is the second leading cause of cancer-related death in women ages 29-39. Despite programs to improve accessibility of cervical cancer screening and overall high screening rates, disparities in routine surveillance have been demonstrated in certain populations, such as victims of intimate partner violence and sexual trauma. One barrier to participating in cervical cancer screening for this population is the office-based visit which necessitates the individual to undress, sit with their legs in stirrups, and undergo speculum examination for specimen collection. This type of visit may cause distress for participants who have experienced sexual violence. HPV self-collection has been studied with favorable outcomes in effectiveness and ease of use. This study evaluates the experience of HPV self-collection among individuals who have experienced sexual trauma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To explore the HPV self-collection experience among individuals with a history of sexual trauma.

OUTLINE:

Participants complete a survey, use an HPV self-collection kit, and attend an interview over 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with a cervix who are eligible for primary HPV testing (age 25 and older) according to national cervical cancer screening guidelines
* Identify themselves as having a history of IPV, sexual abuse, or sexual trauma
* Participants will also need to have access to a smartphone, tablet, or computer with video capability
* English speaking
* Reside in the State of Oregon
* Patients who have participated in prior HPV self-collection study (reference Institutional Review Board [IRB] number- IRB# 23478) will also be eligible to participate in the interview if they meet the remaining eligibility requirements (i.e. history of IPV, sexual abuse, sexual trauma)

Exclusion Criteria:

* Individuals who are not English speaking
* Individuals < 25 years old or no longer eligible/recommended to undergo cervical cancer screening
* Resides outside the state of Oregon
* Adults who are unable to consent or are decisionally impaired
* Individuals without a cervix (i.e. prior hysterectomy)

Min Age: 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Females are individuals with a cervix including women, gender non-forming, non-binary and transgender (trans) persons
Study Population: Individuals with a history of intimate partner violence (IPV), sexual abuse, or sexual trauma and who are eligible for primary HPV based cervical cancer screening.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2022-09-06 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Experience of cervical cancer screening in patients with a history of sexual trauma | Up to 12 months
  Data analysis of interview transcripts will occur concurrent with data collection. The transcripts will be analyzed using Taguette, a qualitative software program. The coding scheme to analyze interview transcripts will be developed through an iterative and reflective process using grounded theory. A comparative, iterative, and interactive method, grounded theory follows a cyclical research process of collecting, analyzing and coding data, memo-writing and theoretical sampling to the point of saturation, where no new ideas, theories or constructs emerge. The research team will thoroughly explore the data and develop a comprehensive list of categories. The categories will be used to identify themes and make connections both between and across interview subjects. Thematic analysis will be basis of the study's findings.
Utility of HPV self-collection among patients with a history of sexual trauma | Up to 12 months
  Data analysis of interview transcripts will occur concurrent with data collection. The transcripts will be analyzed using Taguette, a qualitative software program. The coding scheme to analyze interview transcripts will be developed through an iterative and reflective process using grounded theory. A comparative, iterative, and interactive method, grounded theory follows a cyclical research process of collecting, analyzing and coding data, memo-writing and theoretical sampling to the point of saturation, where no new ideas, theories or constructs emerge. The research team will thoroughly explore the data and develop a comprehensive list of categories. The categories will be used to identify themes and make connections both between and across interview subjects. Thematic analysis will be basis of the study's findings.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda S Bruegl, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States